CLINICAL TRIAL: NCT06759805
Title: eCardiacRehab - a Pragmatic Trial on a Home-based Patient-centered e-Health Programme With Tailored Solutions - Feasibility Study
Brief Title: Electronic Cardiac Rehabilitation (eCardiacRehab) Feasibility Study
Acronym: eCardiacRehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Research Council of Norway (Other); Helse Vest (Other); Helse Fonna (Other); Helse Møre og Romsdal HF (Other Government); Helse Vest IKT (Unknown); Western Norway University of Applied Sciences (Other); Youwell (Unknown); University of Bergen (Other); Østfold University College (Unknown); Norsk råd for digital etikk (Unknown); Helse Førde HF (Unknown); University of Amsterdam (Other); Center for Research on Cardiac Disease in Women (Unknown); Nasjonal kompetansetjeneste Trening som medisin (Unknown); RELIS Vest (Unknown); Norwegian Centre for E-health Research (Unknown); Bergen Municipality (Unknown); Sunnfjord Municipality (Unknown); Sogndal Municipality (Unknown); Masfjorden Municipality (Unknown); The Norwegian Heart and Lung Patient Organization (Unknown); E-helse Vestland (Unknown); Yale University (Other); University of Sydney (Other); University of Cambridge (Other); University of Regina (Other); University of Copenhagen (Other); Linkoeping University (Other Government); Voss Hospital, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 459136; 344337 (Other Grant/Funding Number: Norwegian Research Council); F-12624 (Other Grant/Funding Number: Western Norway Regional Health Authority); R-10930 (Other Grant/Funding Number: Western Norway Regional Health Authority)
Record Dates: First submitted 2024-12-20; First posted 2025-01-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease; Cardiac Rehabilitation; Ethics; Continuity of Patient Care; Older Adults (65 Years and Older); Cost-Benefit Analysis; Adherence, Medication; Adherence, Treatment; Health Literacy; eHealth Literacy; Mental Health; Secondary Prevention of Coronary Heart Disease; Comorbidities; Hypertension; Physical Activity; Women
MeSH Terms: conditions — Coronary Artery Disease; Medication Adherence; Treatment Adherence and Compliance; Psychological Well-Being; Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Usual care
- Intervention group (Other): Digital cardiac rehabilitation
  Interventions: Other: eCardiacRehab

INTERVENTIONS:
Other: eCardiacRehab — Interdisciplinary supervised home-based digital secondary prevention programme (12-week programme) based on the European Society of Cardiology guidelines for cardiac rehabilitation for patients after percutaneous coronary intervention.
  Arms: Intervention group

SUMMARY:
In Norway, more than 11,000 patients undergo percutaneous coronary intervention (PCI) annually. However, a very recent study utilizing registry data show a national average of cardiac rehabilitation (CR) participation of only 14%, despite its proven beneficial effects on readmissions, physical capacity, psychological distress, self-management, and quality of life. CR is strongly recommended in European guidelines. However, uptake is low and is not systematically identifying those in most need of CR. The primary objective of eCardiacRehab is to meet rehabilitation needs of large patient populations regardless of their access to traditional place-based rehabilitation by developing and evaluating the efficacy and cost effectiveness of an interdisciplinary and comprehensive home-based eCardiacRehab programme. eCardiacRehab address patient- and system level challenges in order to increase access to CR. The investigators give particular attention to older patients, women, and those with comorbidities or mental health challenges. Aspects related to continuity of care between specialist and primary care services, health literacy, adherence to treatment, cost effectiveness and ethics are investigated. The investigators will 1) continue to develop the programme with patients, general practitioners, healthcare experts from both specialist and primary care services, and technology developers, 2) develop treatment modules, 3) establish information and communication infrastructure, 4) evaluate the process and efficacy of treatment modules, 5) ensure knowledge development and transfer of competence to the municipalities, and 6) contribute to fulfil the innovation potential for health service and industry partners. eCardiacRehab has the potential to improve interaction and collaboration between primary and secondary care, modernise and digitalise work processes, and develop more coherent and tailored patient pathways. The vision of the home-based eCardiacRehab is to make CR available to all.

ELIGIBILITY:
Inclusion Criteria:

* Adult Norwegian (or Scandinavian) speaking patients (≥ 18 years) who have a Norwegian national identification number,
* With coronary artery disease after percutaneous coronary intervention
* Are living at home and have internet available to them
* Providing signed informed consent

Exclusion Criteria:

* Patients with cognitive impairment that may interfere with the ability to comply with the study protocol
* Severe aortic stenosis
* Severe arrhythmias
* Expected lifetime less than one year as determined by study personnel
* Otherwise clinically unstable
* Not fully revascularized (awaits percutaneous coronary intervention or coronary artery bypass graft surgery)
* Inability to comply with the study protocol due to any physical disability, somatic disease, or mental problems as determined by study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2035-10-30 (Estimated)

PRIMARY OUTCOMES:
The participants' engagement and adherence to the intervention | From start to the end of the programme (12 weeks)
  Based on previous studies, the success criteria will be one login to the website on average once per week, and that 50% of participants will watch some or all the video messages on the website. Usage will be assessed as time spent using the programme, number of logins with start and end time, summary of number of sessions, messages sent, modules completed, and registrations per patient, number of completed questionnaires per patient, and start and end time for all modules in the programme. This will be assessed based on website usage statistics gathered by a website visit tracking system. Further, participants will be asked to report login-errors.
Missing rate | From start to end of programme (12 weeks)
  Acceptability of the secondary and primary outcomes is assessed through response and completion rates. The proportion of missing data in each completed questionnaire at baseline and at the end of the intervention of less than 20% is acceptable.
Attrition rate | From start to the end of programme (12 weeks)
  A success criterion to reduce the threats to validity is an attrition rate of no more than 20%. When possible, the reasons for participants leaving the study are obtained and reported in a study log.

SECONDARY OUTCOMES:
Hospitalization | 180 days hospitalization
  Composite end-point of Emergency Department (ED) contact and home, ED and observation, ED and admission (>24 hours), and death, whichever comes first.
Change in beliefs and perceptions about medicines and treatment | Up to 24 months.
  The Beliefs about Medicines Questionnaire (BMQ) assesses beliefs and perceptions about medicines and treatment. The BMQ comprises two sections: the BMQ-Specific which assesses representations of medication prescribed for personal use and the BMQ-General which assesses beliefs about medicines in general. The two sections of the BMQ can be used in combination or separately. For this study, the BMQ-Specific will be used. Respondents rate 11 items on a 5-point scale ranging from 1 (strongly agree) to 5 (strongly disagree).
Continuity of care | Self-report up to 6 months.
  The Heart Continuity of Care Questionnaire (HCCQ) comprises 33 items covering eight topic areas regarding continuity of care. Respondents rate each item on a 6-point scale ranging from 1 (strongly disagree) to 5 (strongly agree) or 6 (not applicable).
Change in health literacy | Up to 24 months
  The Health literacy questionnaire (HLQ) has nine scale scores that each measure an aspect of the multidimensional construct of health literacy. Each score provides insight into the strengths and limitations of the respondent, but the scores are most powerful when viewed together to show the 'health literacy profile' of the respondent
Anxiety and depression | Up to 24 months
  The Hospital Anxiety and Depression Scale (HADS). The HADS is a fourteen item scale where seven of the items relate to anxiety and seven relate to depression. The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence). The total score is 42 (21 per subscale).
Maximal oxygen consumption (Vo2 max) | Baseline and 12 weeks.
  Maximal oxygen consumption (VO2max) as measured by cardiopulmonary exercise testing (CPET).
Healthcare utilization | Up to 24 months.
  Healthcare utilization will be assessed during follow-up, including patients' use of primary care services (general practitioner visits) and secondary care services (inpatient admissions and outpatient visits). The data source will be nationwide registries. The measurement unit will be mean number of visits.
Healthcare cost | Up to 24 months.
  Health care (associated) costs will be valued using the tariffs of national agreements between the professional associations of medical specialists and the National Health Services. In secondary care, inpatient admissions and outpatient visits will be valued using the tariffs of the national case-mix system of the diagnosis-related groupings (DRG) and the ambulatory grouping system (DAGS). In addition, data will be collected on prescription of medication, which will be valued using the retail price. The data source will be nationwide registries. The measurement unit will be mean costs in Euros.
Change in health status following myocardial infarction | Up to 24 months.
  The Myocardial Infarction Dimensional Assessment Scale (MIDAS) is a PRO measure developed and validated to specifically measure the health status of individuals who have suffered a myocardial infarction. It consist of 7 domains, and is a 35 item scale where respondents rate each item on a 5-point scale ranging from 1 (never) to 5 (always). The function of the MIDAS is to indicate the extent of ill health in each of the seven domains assessed, therefore each dimension is scored separately using a simple scoring methodology.
Change in fatigue | Up to 24 months
  A visual analog scale ranging from 0 (fatigue is not a problem) to 10 (fatigue is a major problem) is used to measure change in fatigue.
Change in eHealth literacy | Up to 24 months
  The eHealth Literacy Scale (Eheals) is an 8-item measure of eHealth literacy developed to measure consumers' combined knowledge, comfort, and perceived skills at finding, evaluating, and applying electronic health information to health problems. Respondents indicate their agreement with statements on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly agree).
Change in medication use | Up to 10 years
  Data related to consumption of prescribed medication are identified through national prescription registries. The registries cover all prescriptions dispensed at pharmacies nationwide. The registries also include information about date of dispensation, quantity and strength dispensed. This will serve as complimentary information to patients' self-reported adherence.
Change in self-reported medication adherence | Up to 24 months
  The my experience of taking medicines (MYMEDS) questionnaire consists of six sections. Section 1: essential contextual information (e.g. the medicines taken). Section 2: overall understanding and satisfaction with medicines (four-point Likert scale (strongly agree, agree, disagree, strongly disagree)). Section 3: areas of anxiety about medicines (e.g. worry that they will cause more harm than good). Section 4: four separate practical concerns associated with medicines taking (e.g. swallowing problems). Section 5: assesses three issues in fitting medicines into patients' daily routine (e.g. relating to forgetfulness or inconvenience). Section 6: asks about adherence to each individual medicine over the past month (five point Likert scale). .
Change in physical and mental dimensions of health | Up to 24 months
  RAND-12 measures physical and mental dimensions of health. The 12 items in the questionnaire correspond to eight principal physical and mental health domains. The 12 items are summarized into two scores, a "Physical Health Summary Measure (PCS-physical component score)" and a "Mental Health Summary Measure (MCS-mental component score)".
Health related quality of life | Up to 24 months
  The HeartQoL questionnaire is a core ischemic heart disease specific health related quality of life (HRQL) questionnaire. The questionnaire comprises 14-items with 10-item physical and 4-item emotional subscales which are scored from 0 (poor HRQL) to 3 (better HRQL) with a global score if needed.
Change in chest pain | Up to 24 months
  The Seattle Angina Questionnaire (SAQ-7) comprises 7 dimensions of coronary artery disease. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Change in self-reported health | Up to 24 months
  EQ-5D-5L is an 5 item (plus a VAS scale) self-report-questionnaire assessing self-reported health. Each question has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Digital health readiness | Up to 24 months
  Responses to the Digital Health Readiness Questionnaire (DHRQ) are scored on a 5-point Likert scale (strongly disagree to strongly agree). The sum of the first 4 domains gives the total score on the DHRQ. The minimum score of the DHRQ is 15, and the maximum score of the DHRQ is 75. Additionally, a fifth domain called digital learnability is assessed.
Change in insomnia | Up to 24 months
  The Minimal Insomnia Symptom Scale (MISS) comprises 3 items assessing major features of insomnia, i.e. difficulties initiating sleep, waking at night and not feeling refreshed by sleep.
Change in sleep | Up to 24 months
  The Sleep Sufficient Index (SSI) comprises 2 items assessing amount of actual and desired sleep.
Medication adherence assessed by therapeutic drug monitoring | Baseline, 3 and 6 months
  Serum levels of cardiac medications (quantified using liquid chromatography with mass spectrometry)
Blood samples | Baseline, 3 and 6 months.
  HbA1c (≤7.0%), lipids, cardiac and inflammation markers(e.g. troponins, natriuretic peptides and CRP).
Change in blood pressure | Up to end of programme
  Blood pressure targets (<120/70 mmHg at nurse visit; <120/70 mmHg at home measurement)
Change in biometrics | Baseline, start and end of programme
  BMI (WHO- classification), visceral fat, muscle mass, body fat.
Change in nicotine status | Up to 24 months
  Self-reported change in nicotine status
Change in self-reported intensity-adjusted minutes | Up to 24 months
  The the physical activity frequency, intensity, and duration (PAFID) questionnaire contains three items on physical activity: (i) frequency [never (0), less than once per week (0.5), once per week (1), 2-3 times per week (2.5), or almost every day (5)]; (ii) duration of each exercise session [<15 min (7.5), 15-29 min (22.5), 30-60 min (45), or over 60 min (75)]; and (iii) intensity [low ('I take it easy, I don't get out of breath or break a sweat'), moderate ('I push myself until I'm out of breath or break into a sweat'), or high ('I practically exhaust myself')]. The number of minutes of physical activity is calculated as the average time spent per session multiplied by the average frequency of exercise per week multiplied by the weighted intensity [low (0.5), moderate (1), and high (2)] based on the values in brackets.
Biosensor data | Throughout the 12-week program
  Biosensor data is collected throughout the 12-week program, and include time spent sedentary and in light-, moderate- and vigorous-intensity physical activity, daily step count, resting/maximal heart rate, sleep time and quality and time and duration of wearing the wearable device.

CONTACTS AND LOCATIONS:
Overall Officials: Tone M Norekvål, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not made available for others according to the Norwegian data protection legislation.

REFERENCES:
- [Background] Brors G, Pettersen TR, Hansen TB, Fridlund B, Holvold LB, Lund H, Norekval TM. Modes of e-Health delivery in secondary prevention programmes for patients with coronary artery disease: a systematic review. BMC Health Serv Res. 2019 Jun 10;19(1):364. doi: 10.1186/s12913-019-4106-1. PMID 31182100
- [Background] Valaker I, Fridlund B, Wentzel-Larsen T, Nordrehaug JE, Rotevatn S, Raholm MB, Norekval TM. Continuity of care and its associations with self-reported health, clinical characteristics and follow-up services after percutaneous coronary intervention. BMC Health Serv Res. 2020 Jan 31;20(1):71. doi: 10.1186/s12913-020-4908-1. PMID 32005235
- [Background] Norekval TM, Allore HG, Bendz B, Bjorvatn C, Borregaard B, Brors G, Deaton C, Falun N, Hadjistavropoulos H, Hansen TB, Igland S, Larsen AI, Palm P, Pettersen TR, Rasmussen TB, Schjott J, Sogaard R, Valaker I, Zwisler AD, Rotevatn S; CONCARD Investigators. Rethinking rehabilitation after percutaneous coronary intervention: a protocol of a multicentre cohort study on continuity of care, health literacy, adherence and costs at all care levels (the CONCARDPCI). BMJ Open. 2020 Feb 12;10(2):e031995. doi: 10.1136/bmjopen-2019-031995. PMID 32054625
- [Background] Norekval TM, Allore HG. Cardiac rehabilitation in older adults: is it just lifestyle? Heart. 2020 Jul;106(14):1035-1037. doi: 10.1136/heartjnl-2019-316497. Epub 2020 Apr 16. No abstract available. PMID 32299827
- [Background] Brors G, Dalen H, Allore H, Deaton C, Fridlund B, Osborne RH, Palm P, Wentzel-Larsen T, Norekval TM; CONCARD investigators. Health Literacy and Risk Factors for Coronary Artery Disease (From the CONCARDPCI Study). Am J Cardiol. 2022 Sep 15;179:22-30. doi: 10.1016/j.amjcard.2022.06.016. Epub 2022 Jul 16. PMID 35853782
- [Background] Brors G, Dalen H, Allore H, Deaton C, Fridlund B, Norman CD, Palm P, Wentzel-Larsen T, Norekval TM. The association of electronic health literacy with behavioural and psychological coronary artery disease risk factors in patients after percutaneous coronary intervention: a 12-month follow-up study. Eur Heart J Digit Health. 2023 Feb 7;4(2):125-135. doi: 10.1093/ehjdh/ztad010. eCollection 2023 Mar. PMID 36974270
- [Background] Instenes I, Fridlund B, Borregaard B, Larsen AI, Allore H, Bendz B, Deaton C, Rotevatn S, Falun N, Norekval TM. 'When age is not a barrier': an explorative study of nonagenarian patients' experiences of undergoing percutaneous coronary intervention. Eur J Cardiovasc Nurs. 2024 Sep 5;23(6):608-617. doi: 10.1093/eurjcn/zvad132. PMID 38243638
- [Background] Hjertvikrem N, Brors G, Instenes I, Helmark C, Pettersen TR, Rotevatn S, Zwisler ADO, Norekval TM; CONCARDPCI Investigators. Use of health services and perceived need for information and follow-up after percutaneous coronary intervention. BMC Res Notes. 2024 Jan 5;17(1):20. doi: 10.1186/s13104-023-06662-y. PMID 38183067
- [Background] Ferrel-Yui D, Candelaria D, Pettersen TR, Gallagher R, Shi W. Uptake and implementation of cardiac telerehabilitation: A systematic review of provider and system barriers and enablers. Int J Med Inform. 2024 Apr;184:105346. doi: 10.1016/j.ijmedinf.2024.105346. Epub 2024 Jan 24. PMID 38281451
- [Background] Norekval TM, Bale M, Bedane HK, Hole T, Ingul CB, Munkhaugen J. Cardiac rehabilitation participation within 6 months of discharge in 37 136 myocardial infarction survivors: a nationwide registry study. Eur J Prev Cardiol. 2024 Nov 18;31(16):1977-1980. doi: 10.1093/eurjpc/zwad350. No abstract available. PMID 37943676
- [Background] Pettersen TR, Schjott J, Allore H, Bendz B, Borregaard B, Fridlund B, Hadjistavropoulos HD, Larsen AI, Nordrehaug JE, Rasmussen TB, Rotevatn S, Valaker I, Wentzel-Larsen T, Norekval TM; CONCARD Investigators. Discharge Information About Adverse Drug Reactions Indicates Lower Self-Reported Adverse Drug Reactions and Fewer Concerns in Patients After Percutaneous Coronary Intervention. Heart Lung Circ. 2024 Mar;33(3):350-361. doi: 10.1016/j.hlc.2023.12.005. Epub 2024 Jan 18. PMID 38238118
- See also: eCardiacRehab study page — https://www.helse-bergen.no/avdelinger/hjarteavdelinga/procard/ehjerterehab